CLINICAL TRIAL: NCT02306681
Title: An International Survey on Hypoglycaemia Among Insulin-treated Patients With Diabetes
Brief Title: A Survey on Low Blod Sugar Among Insulin-treated Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-4177; U1111-1161-9157 (Other: WHO)
Record Dates: First submitted 2014-11-12; First posted 2014-12-03 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SAQ-Self-Assessment Questionnaire
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — This study comprises of a two-part SAQ (Self-Assessment Questionnaire). Paired responses to SAQ1 and SAQ2 will be used to estimate the differences in the frequency of hypoglycaemic episodes between the retrospective and prospective periods.

SUMMARY:
This study is conducted globally. The aim of this study is to describe the proportion of patients with hypoglycaemic episodes and estimate the incidence of various types of hypoglycaemia in the retrospective and prospective periods.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Patient with T1DM or T2DM treated with insulin for more than 12 months
* Male or female patient at least 18 years of age at the time of inclusion in the study

Exclusion Criteria:

* Previous participation in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Illiterate patients and patients otherwise unable to sign the Informed Consent or complete a written survey
* Non-ambulatory patients
* Simultaneous participation in any other clinical study with an investigational product

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients with T1DM (Type 1 Diabetes Mellitus) or T2DM (Type 2 Diabetes Mellitus) treated with insulin for more than 12 months who are 18 years or older, ambulatory, literate, and have signed the Informed Consent form may participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 7315 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2015-05-14 (Actual); Study Completion 2015-05-14 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who experience at least 1 hypoglycaemic episode | During the 4-week prospective observational period

SECONDARY OUTCOMES:
Incidence of any hypoglycaemic episodes | In the 4 weeks before and 4 weeks after the baseline (day 1)
Incidence of hypoglycaemic episodes requiring hospital admission | In the 6 months before and 4 weeks after the baseline (day 1)
Incidence of severe hypoglycaemic episodes | In the 6 months before and 4 weeks after the baseline (day 1)
Incidence of non-severe hypoglycaemic episodes | In the 4 weeks before and 4 weeks after the baseline (day 1)
Incidence of documented symptomatic hypoglycaemic episodes | In the 4 weeks after the baseline visit (day 1)
Incidence of all hypoglycaemic episodes associated with a blood glucose measurement below 3.1 mmol/L (56 mg/dl) irrespective of symptoms | In the 4 weeks following the baseline visit (day 1)
Incidence of hypoglycaemic episodes | Between midnight and 6 a.m. in the 4 weeks before and 4 weeks after the baseline visit (day 1)
Incidence of probable symptomatic hypoglycaemia | In the 4 weeks following the baseline visit (day 1)
Frequency of blood glucose monitoring | Over 1 day
Patient reported fear of hypoglycaemia | Over one day
Patient reported recovery times | One day
Proportion of patients consulting a doctor | Over one day
Proportion of patients increasing calorie intake | Over one day
Proportion of patients avoiding physical exercise | Over one day
Proportion of patients reducing or skipping insulin dose | Over one day
Proportion of patients increasing the number of blood glucose monitoring as a result of fear of hypoglycaemia or hypoglycaemic episodes | Over one day
Proportion of patients taking any sick leave, sick days or short days as a result of hypoglycaemic episodes | Over one day
DSQOLS (Diabetes-Specific Quality-of-Life Scale) scores | Over last 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (8):
- Novo Nordisk Investigational Site, Dhaka, Bangladesh
- Novo Nordisk Investigational Site, Bogotá, Colombia
- Novo Nordisk Investigational Site, Cairo, Egypt
- Novo Nordisk Investigational Site, Manila, Philippines
- Novo Nordisk Investigational Site, Singapore, Singapore
- Novo Nordisk Investigational Site, Pretoria, South Africa
- Novo Nordisk Investigational Site, Ankara, Turkey (Türkiye)
- Novo Nordisk Investigational Site, Ajman, United Arab Emirates

REFERENCES:
- [Background] Pathan F, Goh SY, Rudijanto A, Gadekar A, Jain A, Nicodemus N Jr. Hypoglycaemia among Insulin-Treated Patients with Diabetes: Southeast Asia Cohort of IO HAT Study. J ASEAN Fed Endocr Soc. 2018;33(1):28-36. doi: 10.15605/jafes.033.01.05. Epub 2018 Apr 4. PMID 33442108
- [Result] Emral R, Pathan F, Cortes CAY, El-Hefnawy MH, Goh SY, Gomez AM, Murphy A, Abusnana S, Rudijanto A, Jain A, Ma Z, Mirasol R; IO HAT Investigator Group. Self-reported hypoglycemia in insulin-treated patients with diabetes: Results from an international survey on 7289 patients from nine countries. Diabetes Res Clin Pract. 2017 Dec;134:17-28. doi: 10.1016/j.diabres.2017.07.031. Epub 2017 Aug 9. PMID 28951336
- [Result] Emral R, Tetiker T, Sahin I, Sari R, Kaya A, Yetkin I, Cil SU, Tutuncu NB; IO HAT investigator group. An international survey on hypoglycemia among insulin-treated type I and type II diabetes patients: Turkey cohort of the non-interventional IO HAT study. BMC Endocr Disord. 2018 Feb 13;18(1):9. doi: 10.1186/s12902-018-0238-2. PMID 29433560
- [Result] Pathan MF, Fariduddin M, Nazimuddin K, Mollah AS, Islam Siddiqui MN, Hassan KA, Ferdous HS, Rahman MH, Ashrafuzzaman SM, Sobhan MJ, E-Tanvir Haider MR, Amin MF. The Incidence of Hypoglycemia among Insulin-Treated Patients with Type 1 or Type 2 Diabetes: Bangladeshi Cohort of International Operations-Hypoglycemia Assessment Tool Study. Indian J Endocrinol Metab. 2018 May-Jun;22(3):379-386. doi: 10.4103/ijem.IJEM_545_17. PMID 30090731
- [Derived] Mirasol R, Nicodemus N Jr, Jain A, Gadekar AV, Yu-Gan S. Self-Reported Hypoglycemia in Insulin-Treated Patients with Diabetes: Results from the Philippine Cohort of the International Operations Hypoglycemia Assessment Tool (IO HAT) Study. J ASEAN Fed Endocr Soc. 2018;33(1):12-21. doi: 10.15605/jafes.033.01.03. Epub 2018 Apr 3. PMID 33442106
- [Derived] Gomez AM, Chica LG, Burbano AF, Vasquez EM, Escobar JA, Arias PM, Molina DI. Survey on hypoglycemia among insulin-treated patients with diabetes: The Colombian International Operations Hypoglycemia Assessment Tool population. Biomedica. 2019 Sep 1;39(3):576-586. doi: 10.7705/biomedica.4365. PMID 31584770
- [Derived] Rudijanto A, Saraswati MR, Yunir E, Kumala P, Puteri HH, Mandang VV. Indonesia Cohort of IO HAT Study to Evaluate Diabetes Management, Control, and Complications in Retrospective and Prospective Periods Among Insulin-Treated Patients with Type 1 and Type 2 Diabetes. Acta Med Indones. 2018 Jan;50(1):26-37. PMID 29686173
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com